CLINICAL TRIAL: NCT00594776
Title: Vascular CT Assessment of Structural Autograft and Allograft Healing
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Eddie Schwarz, Professor, University of Rochester
Other Study IDs: 15198; P50AR054041 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Bone Tumors
Keywords: Cone Beam CT; CBCT; Bone Tumors; Autographs; Allographs
MeSH Terms: conditions — Bone Neoplasms | interventions — Tomography, Spiral Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who have received a structrual allograft or vascularized fibular autograft surgery to reconstruct their tibia, femur, ulna/radius or humerus for treatment of a bone tumor.
  Interventions: Device: Cone Beam CT Scan

INTERVENTIONS:
Device: Cone Beam CT Scan — The Cone Beam Computerized Tomographic (CBCT) device utilizes computerized tomographic technology, a special digital imaging plate and a computer to create a three-dimensional image. The special imaging plate and software allow for small details to be imaged without tissue overlap.

SUMMARY:
The purpose of this study is to determine the ability of a cone beam CT to measure bone healing.

DETAILED DESCRIPTION:
The purpose of this study is to investigate quantitative vascular cone beam CT(CBCT) in a clinical pilot of patients that have received a structural allograft for bone cancer or a vascularized structural autograft for bone cancer or traumatic injury. Development of a minimally invasive, longitudinal outcome measure to quantify intramedullary vascular volume and cortical bone volume of structural allografts in patients is required to translate "revitalizing" structural allograft in clinical trials. Our novel vascular CBCT will be able to demonstrate the significant differences between vascularized fibular autografts vs. structural allografts in patients that will undergo structural grafting. These data will be used to devise a power calculation for a definitive clinical trial to evaluate the efficacy of the revitalizing allograft.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* all races will be included
* autograft or allograft of long bone as part of treatment for bone tumor

Exclusion Criteria:

* pregnancy
* patients with a history of IV contrast reactions
* contraindication to use of epinephrine or diphenhydramine
* hypertyroidism or history of sensitivity to iodine
* kidney disease (abnormal urinalysis or calculaged GFR) or poor hydration due to poor intake or other causes

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are recruited from the general practice of 3 of our investigators. Patients will have received an structural allograft or vascularized autograft for the treatment of bone cancer.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in intramedullary vascular volume and new bone growth based on CBCT | 2, 8 & 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Schwarz, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States